CLINICAL TRIAL: NCT07195123
Title: Evaluation of the SMART IBD App Digital Therapeutic Tool for Pediatric Inflammatory Bowel Disease
Brief Title: Evaluation of the SMART IBD App in Pediatric IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMART-IBD R21 RCT
Record Dates: First submitted 2025-09-17; First posted 2025-09-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease (IBD); IBD (Inflammatory Bowel Disease); IBD - Inflammatory Bowel Disease; Ulcerative Colitis (UC); Indeterminate Colitis; Crohn Disease (CD); IBD
Keywords: IBD; Inflammatory Bowel Disease; Ulcerative Colitis; Indeterminate Colitis; Crohns Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study PI, statistician, co-investigators, and all personnel who are involved in endpoint analyses will be blinded. Only study coordinators will have access to the assignment of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-IBD App (Experimental): The SMART-IBD app consists of educational content, medication reminders, and monthly app engagement challenges. App users will participate in 5 monthly challenges that focus on topics such as adherence, sleep, and diary usage. Participants in this arm will complete one month of run-in diaries, a baseline assessment, 5 months of intervention, including daily symptom diaries, and a post-treatment assessment.
  Interventions: Behavioral: SMART-IBD
- Attention Control (No Intervention): Participants in this arm will not receive any intervention content. Participants in this arm will complete one month of run-in diaries, a baseline assessment, 5 months of daily symptom diaries, and a post-treatment assessment.

INTERVENTIONS:
Behavioral: SMART-IBD — Daily medication and diary completion reminders are provided to participants. Additional psychoeducational content regarding self-management skills will be provided in-app.
  Arms: SMART-IBD App

SUMMARY:
The objective of this trial is to test whether a smartphone app, SMART-IBD, is effective in improving medication adherence and self-management skills in adolescents with IBD. The investigators will conduct a randomized control trial to compare 35 youth (ages 13-17) with IBD using an app that contains daily symptom diaries, education content, medication reminders, as well as monthly engagement challenges to 35 youth in an attention control group that will complete daily diaries. The length of the intervention will include one month of baseline symptom and adherence collection, a baseline assessment, 5 months of intervention, and a post-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of IBD (Crohn's Disease, ulcerative colitis, or indeterminate colitis)
* Prescribed at least one daily or weekly medication for treatment of IBD
* <86% adherence to prescribed medication
* Access to internet via Wi-Fi or data plan and access to smartphone
* English fluency for patient and caregiver

Exclusion Criteria:

* Diagnosis of pervasive developmental disorder in patient or caregiver as determined by medical chart review
* Diagnosis of serious mental illness (e.g., schizophrenia) in patient or caregiver as determined by medical chart review

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 6 months
  Medication adherence will be measured by daily responses by participants to prompts in the SMART IBD app regarding whether each dose was taken for each medication. A mean adherence score will be calculated across medications for each participant for the 28 day periods at baseline and post-treatment.

SECONDARY OUTCOMES:
Disease Activity | 6 months
  PROs will be collected regarding composite disease activity comprised of fecal calprotectin, stool frequency, and rectal bleeding for ulcerative colitis and fecal calprotectin, stool frequency, and abdominal pain for Crohn's. Stool samples collected at baseline and post-assessment will also be utilized to assess diseases activity.
Sleep Duration | 6 months
  Sleep duration will be assessed via the SMART IBD App diary on a scale of 0-18 hours or more with half hour increments. Participants in both arms will report sleep duration via the diary.
Stress | 6 months
  Stress will be assessed via the SMART IBD App diary on a scale of 0-10, where 0 is no stress and 10 is highest stress. Participants in both arms will report stress via the diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States